CLINICAL TRIAL: NCT05261984
Title: Investigating the Anabolic Response to Resistance Exercise After Critical Illness: The ARTIST-2 Non-Randomized Controlled Trial
Brief Title: Investigating the Anabolic Response to Resistance Exercise After Critical Illness (ARTIST-2)
Acronym: ARTIST-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Martin Sundstrom Rehal, Principal Investigator, Karolinska University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K 2022-1113
Record Dates: First submitted 2022-02-20; First posted 2022-03-02 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Critical Illness; Muscle Loss
Keywords: Resistance exercise; Muscle protein; Anabolic resistance
MeSH Terms: conditions — Critical Illness; Muscular Atrophy | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Former ICU patients (Experimental): Research subjects with a prior history of ICU treatment within six months.
  Interventions: Procedure: Resistance exercise; Dietary Supplement: Oral protein supplementation
- Age- and sex-matched control group (Active Comparator): Research subjects without a prior history of ICU treatment within the last 30 years, age- and sex-matched in a 1:2 ratio to the experimental arm.
  Interventions: Procedure: Resistance exercise; Dietary Supplement: Oral protein supplementation

INTERVENTIONS:
Procedure: Resistance exercise — Knee extensions in flywheel inertia machine in four sets of 10 repetitions.
Dietary Supplement: Oral protein supplementation — 24 grams of hydrolyzed whey protein.

SUMMARY:
ICU survivors often suffer from long-term functional disability. An attenuated response to physical exercise in skeletal muscle after critical illness may contribute to persisting weakness.

The aim of this study is to investigate the effects of resistance exercise on muscle protein synthesis in former ICU patients. The investigators hypothesize that study subjects recovering from critical illness have an impaired anabolic response to resistance exercise after ICU stay as compared to non-critically ill controls.

DETAILED DESCRIPTION:
Background

The debilitating impact of critical illness has been recognized for several decades. Disability related to intensive care is now described as a syndrome called ICU-acquired weakness (ICUAW). ICUAW affects up to 70% of ICU patients and is most common with higher illness severity. Patients that develop ICUAW require longer hospitalization and have a higher risk of death. Weakness may persists for several years in ICU survivors. It has significant long-term consequences, and is associated with increased health care costs, delayed return to work, and overall poor quality of life.

Muscle atrophy is a major contributor to ICUAW. Critical illness is associated with a rapid loss of skeletal muscle, induced by catabolic signals from proinflammatory cytokines and hormones. The ability to regain lost muscle mass during convalescence may also be impaired. In a small observational study, muscle atrophy resolved only in a minority of ICU survivors at six months after ICU discharge.

Studies in exercise physiology have demonstrated that resistance training and amino acid ingestion have synergistic effects on muscle protein synthesis in healthy subjects. It is therefore an appealing therapy to reconstitute muscle mass after critical illness. Despite several clinical trials, there is equipoise regarding the efficacy of exercise in improving physical function in-ICU after ICU discharge. These mixed signals are unsurprising given the heterogeneous causes of ICUAW.

Only a few studies in this field have examined muscle architecture or cellular signaling in response to training. However, the gold standard in determining the anabolic response to exercise is to directly measure the effects on protein synthesis and breakdown. There is still no published research using this methodology to assess the effects of exercise interventions in former ICU patients. To understand the role of physical exercise in regaining lost muscle mass, the investigators plan to investigate the anabolic effects to resistance training after critical illness.

Aim and hypothesis

The aim of this study is to determine the anabolic response to resistance exercise after critical illness. The investigators hypothesize that study subjects recovering from critical illness have an impaired anabolic response to resistance exercise after ICU stay as compared to non-critically ill controls.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥18 years) previously admitted to an ICU at Karolinska University Hospital for ≥3 days and discharged alive from hospital

   OR
2. Adult (≥18 years) without a history of ICU admission (control group)

Exclusion Criteria:

1. Not able to provide informed consent
2. >6 months since ICU discharge*
3. Warfarin or dual antiplatelet therapy
4. Clinically significant inherited or acquired disorder of hemostasis
5. Lower-limb amputee
6. Lower-limb atherosclerotic disease with critical ischemia.
7. Recent fracture in lower limbs or significant osteoarthritis limiting movement in knee or hip joint
8. Metastatic cancer or active hematological malignancy
9. Inherited disorder of amino acid metabolism.
10. Chronic muscle, neuromuscular or neurologic disease with prior documentation of clinically significant lower-limb involvement
11. Pregnancy
12. Single organ failure not requiring invasive mechanical ventilation during ICU stay*
13. Intubated only for airway protection with no other organ failure(s) during ICU stay*
14. Planned postoperative care in ICU after elective cardiothoracic surgery*

Exclusion criteria marked with asterisk only apply to former ICU patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Muscle protein fractional synthetic rate | 150 minutes post-exercise.
  The difference between the experimental and active comparator group in muscle protein fractional synthetic rate.

SECONDARY OUTCOMES:
Gene expression | 150 minutes post-exercise.
  The difference between the experimental and active comparator group in gene expression (mRNA) in skeletal muscle, assessed by RNA sequencing.
Signaling pathways | 150 minutes post-exercise.
  The difference between the experimental and active comparator group in the activity of major anabolic/catabolic signalining pathways in skeletal muscle, assessed by western blot.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Sundström Rehal, MD PhD, Principal Investigator — Karolinska University Hospital; Olav Rooyackers, PhD, Study Chair — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Huddinge, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Batt J, Herridge MS, Dos Santos CC. From skeletal muscle weakness to functional outcomes following critical illness: a translational biology perspective. Thorax. 2019 Nov;74(11):1091-1098. doi: 10.1136/thoraxjnl-2016-208312. Epub 2019 Aug 20. PMID 31431489
- [Background] Herridge MS, Tansey CM, Matte A, Tomlinson G, Diaz-Granados N, Cooper A, Guest CB, Mazer CD, Mehta S, Stewart TE, Kudlow P, Cook D, Slutsky AS, Cheung AM; Canadian Critical Care Trials Group. Functional disability 5 years after acute respiratory distress syndrome. N Engl J Med. 2011 Apr 7;364(14):1293-304. doi: 10.1056/NEJMoa1011802. PMID 21470008
- [Background] Plank LD, Connolly AB, Hill GL. Sequential changes in the metabolic response in severely septic patients during the first 23 days after the onset of peritonitis. Ann Surg. 1998 Aug;228(2):146-58. doi: 10.1097/00000658-199808000-00002. PMID 9712558
- [Background] Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, Hopkinson NS, Phadke R, Dew T, Sidhu PS, Velloso C, Seymour J, Agley CC, Selby A, Limb M, Edwards LM, Smith K, Rowlerson A, Rennie MJ, Moxham J, Harridge SD, Hart N, Montgomery HE. Acute skeletal muscle wasting in critical illness. JAMA. 2013 Oct 16;310(15):1591-600. doi: 10.1001/jama.2013.278481. PMID 24108501
- [Background] Wolfe RR. Skeletal muscle protein metabolism and resistance exercise. J Nutr. 2006 Feb;136(2):525S-528S. doi: 10.1093/jn/136.2.525S. PMID 16424140
- [Background] Doiron KA, Hoffmann TC, Beller EM. Early intervention (mobilization or active exercise) for critically ill adults in the intensive care unit. Cochrane Database Syst Rev. 2018 Mar 27;3(3):CD010754. doi: 10.1002/14651858.CD010754.pub2. PMID 29582429
- [Background] Connolly B, Salisbury L, O'Neill B, Geneen L, Douiri A, Grocott MP, Hart N, Walsh TS, Blackwood B; ERACIP Group. Exercise rehabilitation following intensive care unit discharge for recovery from critical illness. Cochrane Database Syst Rev. 2015 Jun 22;2015(6):CD008632. doi: 10.1002/14651858.CD008632.pub2. PMID 26098746
- [Background] Fossat G, Baudin F, Courtes L, Bobet S, Dupont A, Bretagnol A, Benzekri-Lefevre D, Kamel T, Muller G, Bercault N, Barbier F, Runge I, Nay MA, Skarzynski M, Mathonnet A, Boulain T. Effect of In-Bed Leg Cycling and Electrical Stimulation of the Quadriceps on Global Muscle Strength in Critically Ill Adults: A Randomized Clinical Trial. JAMA. 2018 Jul 24;320(4):368-378. doi: 10.1001/jama.2018.9592. PMID 30043066
- [Background] Hickmann CE, Castanares-Zapatero D, Deldicque L, Van den Bergh P, Caty G, Robert A, Roeseler J, Francaux M, Laterre PF. Impact of Very Early Physical Therapy During Septic Shock on Skeletal Muscle: A Randomized Controlled Trial. Crit Care Med. 2018 Sep;46(9):1436-1443. doi: 10.1097/CCM.0000000000003263. PMID 29957714

DOCUMENTS (1):
  • Study Protocol (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/84/NCT05261984/Prot_000.pdf